CLINICAL TRIAL: NCT02923544
Title: Pilot Trial of YUMI Uterine Manipulator
Brief Title: Trial of YUMI Uterine Manipulator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-1397
Record Dates: First submitted 2016-10-03; First posted 2016-10-04 (Estimated); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Gynecologic Condition; Scheduled for a Total Laparoscopic or Robotic-assisted Hysterectomy
Keywords: Uterine Manipulator; Yukio's Uterine Manipulating Instrument (YUMI); 16-1397

ARMS (1):
- total laparoscopic or robotic-assisted hysterectomy (Experimental): The YUMI manipulator will be placed at the start of each case. During the surgery, the surgeon will track any intraoperative complications. The surgeon fellow will also note the feasibility of placing the uterine manipulator.After surgery, the surgeon will complete the product evaluation form.
  Interventions: Procedure: YUMI manipulator

INTERVENTIONS:
Procedure: YUMI manipulator
  Other Names: Yukio's Uterine Manipulating Instrument

SUMMARY:
The purpose of this study is to test the feasibility and safety of using a new device called Yukio's Uterine Manipulating Instrument (YUMI). The YUMI is a type of uterine manipulator. It is a reusable metal device designed to be simple and study. It is also adjustable in size which makes it easy for surgeons to use. It will be placed at the beginning of the surgery and removed at the end. This study will allow the researchers to find out if the surgeons find the YUMI effective and easy to use. It will also allow the researchers to see if the device is safe. This is the first time that the YUMI is being used in humans.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be scheduled for a total laparoscopic or robotic-assisted hysterectomy for a gynecologic condition
* Participants must be 18 years of age or older

Exclusion Criteria:

* Participant is not eligible if the surgeon does not plan to use a uterine manipulator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
number of successfully placed Uterine Manipulator | 1 year
  The YUMI manipulator will be considered successfully placed when the device is inserted into the uterus and secured in place to hold for the duration of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Yukio Sonoda, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent and Follow-Up only), Basking Ridge, New Jersey
  - Memoral Sloan Kettering Monmouth (Consent and Follow-Up only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent and Follow-Up only), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent and Follow-Up only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent and Follow-Up only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent and Follow-Up only), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/